CLINICAL TRIAL: NCT01737619
Title: Prospective Evaluation of Lymph Node Metastasis at the Time of Surgical Staging for High Risk Endometrial Cancer
Brief Title: PET/CT and Lymph Node Mapping in Finding Lymph Node Metastasis in Patients With High-Risk Endometrial Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-0623; NCI-2015-01898 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0623 (Other: M D Anderson Cancer Center); P50CA098258 (NIH)
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Clear Cell Adenocarcinoma; Endometrial Mixed Adenocarcinoma; Endometrial Serous Adenocarcinoma; Grade 3 Endometrial Endometrioid Adenocarcinoma; Malignant Mixed Mesodermal (Mullerian) Tumor
MeSH Terms: conditions — Mixed Tumor, Mesodermal | interventions — Indocyanine Green; Lymph Node Excision; Magnetic Resonance Spectroscopy

ARMS (1):
- Diagnostic (PET/CT, lymph node mapping) (Experimental): Patients undergo PET/CT prior to surgery. Patients then undergo intraoperative lymph node mapping with indocyanine green solution, given via superficial and deep cervical injection during full lymphadenectomy.
  Interventions: Procedure: Computed Tomography; Drug: Indocyanine Green Solution; Other: Laboratory Biomarker Analysis; Procedure: Lymph Node Mapping; Procedure: Lymphadenectomy; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Drug: Indocyanine Green Solution — Given via superficial and deep cervical injection
  Other Names: IC-GREEN; ICG Solution
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Lymph Node Mapping — Undergo lymph node mapping
  Other Names: lymphatic mapping
Procedure: Lymphadenectomy — Undergo full lymphadenectomy
  Other Names: excision of the lymph node; Lymph Node Dissection; lymph node excision
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This clinical trial studies positron emission tomography (PET)/computed tomography (CT) and lymph node mapping in finding lymph node metastasis in patients with endometrial cancer that is at high risk of spreading. A PET/CT scan is a procedure that combines the pictures from a PET scan and a CT scan, which are taken at the same time from the same machine. The combined scans give more detailed pictures of areas inside the body than either scan gives by itself. Lymph node mapping uses a radioactive dye, called indocyanine green solution, to identify lymph nodes that may contain cancer cells. PET/CT and sentinel lymph node mapping may be better ways than surgery to identify cancer in the lymph nodes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the false negative rate of PET/CT and/or sentinel lymph node mapping in the detection of positive lymph nodes in women with high risk endometrial cancers.

SECONDARY OBJECTIVES:

I. To estimate the sensitivity, specificity, positive predictive value, and negative predictive value of PET/CT and/or sentinel lymph node mapping in the detection of positive lymph nodes in women with high risk endometrial cancer.

II. To determine if a molecular panel of estrogen-induced genes that we have previously identified from retrospective studies correlate with extra-uterine spread including lymph node metastasis at the time of surgical staging for endometrial cancer.

III. To prospectively identify patterns of lymphatic spread of endometrial cancer.

IV. To correlate cancer antigen 125 (CA-125) and WAP four-disulfide core domain 2 (HE4) levels with disease metastasis at the time of surgical staging and to explore the use of other serum biomarkers to predict recurrence.

V. To prospectively collect morbidity and mortality data related to performing lymph node dissection including intra-operative and postoperative complications.

VI. To determine whether metabolic parameters of the primary endometrial tumor on PET including tumor intensity (maximum standard uptake value [SUV] and peak SUV), metabolic tumor volume (obtained at a threshold of 40% of maximum and at a threshold of SUV=3), and total lesion glycolysis (expressed average SUV over the metabolic tumor volume) are predictive of locoregional or metastatic spread, and whether these parameters correlate with CA-125 and HE4 levels.

OUTLINE:

Patients undergo PET/CT prior to surgery. Patients then undergo intraoperative lymph node mapping with indocyanine green solution, given via superficial and deep cervical injection during full lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high grade endometrial cancer including grade 3 endometroid, serous, clear cell, malignant mixed Mullerian tumor (MMMT) or any mixed tumor containing one of these cell types
* Patients with a grade 1/2 tumors and evidence of deep myometrial invasion or cervical involvement on preoperative imaging or physical exam
* Candidate for surgery
* No evidence of peritoneal disease on preoperative imaging
* Negative pregnancy test if of child-bearing age
* No preoperative treatment for endometrial cancer including radiation or chemotherapy
* Previous hormonal therapy is allowed

Exclusion Criteria:

* Medical co-morbidities making surgery unsafe, as determined by the primary treating physician
* Any contraindications to PET/CT or lymph node mapping (inability to control serum glucose to a value of =< 200 mg/dl for fludeoxyglucose F-18 [FDG]-PET/CT)
* Does not meet histologic criteria
* Evidence of peritoneal or distant metastasis on preoperative imaging
* Baseline creatinine (necessary for imaging studies)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-04-03 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Soliman, Principal Investigator — M.D. Anderson Cancer Center
Locations (7):
- United States (7):
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - MD Anderson Regional Care Center-Katy, Houston, Texas
  - MD Anderson Regional Care Center-Bay Area, Nassau Bay, Texas
  - MD Anderson Regional Care Center-Sugar Land, Sugar Land, Texas
  - MD Anderson Regional Care Center-The Woodlands, The Woodlands, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was active from April 2013 until May 2016 and all recruitments were done in a medical clinic setting.
Groups:
- Sentinel Node Mapping: Pre-op PET/CT scan followed by intraoperative sentinel lymph node mapping and biopsy then complete pelvic and para-aortic lymphadenectomy
Period: Overall Study
Arm/Group | Sentinel Node Mapping
Started | 101
Completed | 101
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sentinel Node Mapping
Number analyzed (Participants) | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 37
Age, Continuous [Mean (Full Range); unit: years] | 62 [29 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 63
  More than one race | 0
  Unknown or Not Reported | 19
Region of Enrollment [Number; unit: participants]
  United States | 101

OUTCOME MEASURES:

1. Primary Outcome: False Negative Rate of PET/CT Verses Sentinel Lymph Node Mapping in the Detection of Positive Lymph Nodes in Women With High Risk Endometrial Cancers.
Time Frame: 36 months
Measure: Number; unit: percentage
Arm/Group | Sentinel Node Mapping
Number analyzed (Participants) | 101
percentage
  , sensitivity of sentinel lymph node mapping | 95
  false negative rate | 5
  false negative predictive value | 1.4

2. Secondary Outcome: False Negative Rate and False Negative Predictive Values of Lymphatic Spread of Endometrial Spread of Endometrial Lymph Nodes From a PET/CT Versus Lymphatic Mapping Procedure
Time Frame: 36 months
Measure: Number; unit: percentage
Arm/Group | Sentinel Node Mapping
Number analyzed (Participants) | 101
percentage
  false negative rate | 4.3
  false negative predictive value | 1.4

3. Secondary Outcome: Mortality Rate of Patients Undergoing Lymph Node Dissection Including Intra-operative and Postoperative Complications
Description: Mortality percentage of patients following the lymph node mapping procedure and postoperative complications.
Time Frame: 36 months
Measure: Number; unit: percentage of participants
Arm/Group | Sentinel Node Mapping
Number analyzed (Participants) | 101
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: 36 months
Description: NCI CTCAE Version 4.03
Arm/Group | Sentinel Node Mapping
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 0/101
Other Adverse Events (participants affected / at risk) | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT01737619/Prot_SAP_000.pdf